CLINICAL TRIAL: NCT06473324
Title: Association Between Preoperative Persistent Hyperglycemia and Postoperative Delirium in Geriatric Hip Fracture Patients
Brief Title: Association Between Preoperative Hyperglycemia and Postoperative Delirium in Geriatric Hip Fracture Patients
Status: Completed | Type: Observational
Sponsor: Wenbo Ding (Other)
Responsible Party: Sponsor-Investigator, Wenbo Ding, Professor, Dandong Central Hospital
Organization: Dandong Central Hospital (Other)
Other Study IDs: DDZX-20231121
Record Dates: First submitted 2024-06-18; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Delirium; Hip Fractures; Hyperglycemia
MeSH Terms: conditions — Emergence Delirium; Hip Fractures; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hyperglycaemia group: Blood glucose level ≥ 6.1 mmol/L
- hypoglycaemic group: Blood glucose level < 6.1 mmol/L

SUMMARY:
This retrospective study aims to collect electronic medical record data from Dandong central hospital spanning from January 2013 to November 2023. The collected data does not contain any personally identifiable information or breach privacy. Additionally, this study design does not involve active intervention measures or patient recruitment. The research aims to investigate the correlation between preoperative blood glucose levels in elderly hip fracture patients and postoperative delirium.

DETAILED DESCRIPTION:
A retrospective observational study is planned to explore specific phenomena or associations using electronic medical record data. The collected data does not contain any personally identifiable information or compromise privacy. Additionally, this study design does not involve active intervention measures or patient recruitment. The study data is sourced from the electronic medical record system of hospitalized patients and has received approval from the hospital's research center, with ongoing supervision by the hospital's ethics committee. The study aims to investigate the correlation between preoperative blood glucose levels in hip fracture patients and postoperative complications.

The retrospective study aims to collect electronic medical record data spanning from January 2013 to November 2023. The data collection process is consistently monitored and verified by the hospital's ethics committee. Throughout the study, adherence to the ethical principles outlined in the 1964 Helsinki Declaration is ensured, and institutional review board (IRB) approval has been obtained for all aspects of the research.

The study aims to provide valuable evidence-based medicine for clinical practitioners by examining the relationship between preoperative persistent hyperglycemia in elderly hip fracture patients and postoperative delirium. Furthermore, it seeks to offer clinical insights for early identification and intervention management of high-risk postoperative delirium patients (POD).

ELIGIBILITY:
Inclusion Criteria:

1) Patients who have undergone surgical treatment for hip fractures.

Exclusion Criteria:

1. Multiple or pathological hip fractures.
2. Emergent surgery.
3. Age below 60 years.
4. Incomplete electronic medical records or preoperative blood glucose levels were assessed fewer than two times.
5. Presence of neurological and psychiatric disorders, except dementia.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 2,031 electronic medical records were gathered. Following stringent inclusion and exclusion criteria, a retrospective cohort study was conducted on 1,440 patients with hip fracture. Among them, 783 patients (54.4%) exhibited preoperative persistent hyperglycemia (serum glucose levels ≥ 6.1 mmol/L on multiple occasions), while 275 patients (19.1%) experienced postoperative delirium. The average age of the included geriatric hip fracture patients was 74.7 ± 9.8 years, with males comprising 39.7% of the sample.
Sampling Method: Non-Probability Sample
Enrollment: 2031 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Postoperative Delirium | up to 2 months
  Postoperative Delirium (POD) manifests as acute cognitive dysfunction and consciousness disorder, characterized by changes in attention or consciousness that cannot be attributed to pre-existing cognitive impairments. Typical symptoms include hallucinations, delusions, agitated behavior, disordered speech, decreased attention, confusion, unclear consciousness, and disrupted sleep-wake cycles. Moreover, POD typically occurs within the first five days after surgery, particularly within the initial 48 hours, and exhibits significant fluctuations.

CONTACTS AND LOCATIONS:
Locations (1):
- Dandong Central Hospital, Dandong, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang W, Zhang Y, Yao W, Tang W, Li Y, Sun H, Ding W. Association between preoperative persistent hyperglycemia and postoperative delirium in geriatric hip fracture patients. BMC Geriatr. 2024 Jul 8;24(1):585. doi: 10.1186/s12877-024-05192-x. PMID 38977983